CLINICAL TRIAL: NCT05212441
Title: ADJUNCTIVE EFFECT OF LIGHT EMITTING DIODE ON HAND GRIP STRENGTH IN BURN PATIENTS: A Randomized Controlled Trial
Brief Title: ADJUNCTIVE EFFECT OF LIGHT EMITTING DIODE ON HAND GRIP STRENGTH IN BURN PATIENTS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy Ali Hassan ElMeligie, Principal investigator, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LEDHB2122
Record Dates: First submitted 2022-01-15; First posted 2022-01-28 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Burns; Hand Burn; Hand Grasp; Hand Injuries
MeSH Terms: conditions — Burns; Hand Injuries | interventions — Patient Positioning; Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (LED group) (Experimental): This group includes 30 burned patients who will receive LED therapy in addition to their physical therapy program (splinting, stretching ex., strengthening ex. and ROM ex.) and medical treatment.
  Interventions: Device: Light emitting diode therapy (LED therapy); Behavioral: Patient/family education program (Home program); Procedure: Positioning & Splinting; Other: Therapeutic Exercises
- Group B (Control group) (Active Comparator): This group includes 30 burned patients who will receive their physical therapy program (splinting, stretching ex., strengthening ex. and ROM ex.) and medical treatment.
  Interventions: Behavioral: Patient/family education program (Home program); Procedure: Positioning & Splinting; Other: Therapeutic Exercises

INTERVENTIONS:
Device: Light emitting diode therapy (LED therapy) — The patient's forearm is positioned on table with palm facuing upward during the therapy. For LEDT, the center of the light spot located at approximately 50% of landmark line from the medial epicondyle to the styloid process of the ulna, which is the center belly of ﬂexor digitorum superﬁcialis. The subject's forearm maintained in the rest state without moving during the therapy. LED is performed before exercise.
  Arms: Group A (LED group)
Behavioral: Patient/family education program (Home program) — Patients and their families will instructed to learn the anti contracture positioning/splinting, scar massage and exercises program, application of the custom garments and inserts, and functional training to perform them on their own at home. Written and illustrative instructions and reciprocal demonstration sessions will be provided to the children and their families to ensure successful acquisition and delivery of rehabilitation skills at home program. The therapist will be reported about compliance with the home program every couple of days
Procedure: Positioning & Splinting — The wrist joint is splinted at 30 hyperextension, the MCP joint in 90 of flexion, the IP joints in extension, and the thumb in abduction. The webs of fingers kept in abduction. The hands are elevated above the level of the heart to minimize post-burn edema.
  Splinting: Splints are tailored to help to maintain the functional or anti-contracture position of the injured body parts.The intervals for monitoring vary from once every hour to once every 4-6 hours, depending on types of splints and skin conditions. It is described as 10 hours on and two hours off. When the splint is taken off, active and/or passive ROM should be carried out.
Other: Therapeutic Exercises — 1. Passive ROM (PROM).
  2. Active ROM (AROM) & Active-assistive ROM (AAROM): The exercise will focus on extending the wrist to 45 degrees, flexing the MCP joints to 90 degrees and keeping the IP joints in full extension, while maintaining a thumb web space. The exercises will performed in the following sequences; (1) MCP joints flexion and extension with the wrist in neutral or slight extension and the IP joints in neutral position. (2) IP joints flexion to only 30-40 degrees with the wrist stabilized in the neutral or slight extension, while the MCP joints held in full extension, (3) thumb and fingers abduction and adduction, and (4) thumb opposition (tip of the thumb to tip of the small finger). Each exercise was performed for 8-10 repetition, daily, for 6 days/week.
  3. Stretching exercises: A low-load (low-intensity), long-duration stretch
  4. Strengthening exercises: done in static mode initially and progress to dynamic strengthening using elastic bands.

SUMMARY:
This study will be done to evaluate effect of applying LED before hand exercise on hand grip strength. Sixty male patients with subacute partial thickness burn of hand will be randomly allocated into two equal groups of 30 patients. The following equipment and tools will be used

Measurement equipments:

* For total active motion of fingers (TAM): Goniometer.
* For hand grip strength: Hand grip dynamometer.

Therapeutic equipment:

Light emitting diode therapy (LED) device.

ELIGIBILITY:
Inclusion Criteria:

The subject selection will be according to the following criteria:

* Burn caused by thermal injury (flame or scald) with involvement of the wrist and hand and other parts of the body not including shoulder and elbow.
* Age range between 20-35 years.
* Male gender.
* Subacute Partial-thickness burn " From 3rd day of burn".
* Recent discharge of in patient acute care, spontaneous healing.
* All patients enrolled to the study will have their informed consent.

Exclusion Criteria:

The potential participants will be excluded if they meet one of the following criteria:

* Cardiac diseases.
* Perception of persistent respiratory problem related to a previous inhalation injury
* Signs of burn infection (i.e., unclear fluid oozing from the wound, increased pain, expanded redness and swelling)
* Exposed tendons.
* Nerve, muscle injury.
* Scar contracture of hand.
* Cognitive disorders.
* Presence of fractures.
* Patients who suffer from skin diseases, diabetes, varicose veins, and peripheral vascular diseases.
* Patients with life threatening disorders as renal failure, myocardial infarction or other similar diseases will be excluded from the study.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-02-25 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-10 (Estimated)

PRIMARY OUTCOMES:
Changes in Total active ROM from baseline to 6 weeks posttreatment | baseline and 6 weeks posttreatment
  Total active ROM is the sum of the active metacarpophalangeal (MP), proximal interphalangeal (PIP), and distal interphalangeal (DIP) arc of motion in degrees of an individual digit. The measurement will be performed via a hand-held finger goniometer
Changes in hand grip strength from baseline to 6 weeks posttreatment | baseline and 6 weeks posttreatment
  A calibrated hydraulic JAMAR (Model: 5030J1, Sammons Preston Rolyan, Chicago, USA), analogue hand-grip dynamometer will be used to measure grip strength. The device provides 1 kg increments on the measurement dial which faces the assessor as mentioned by Clifford et al., 2013.

CONTACTS AND LOCATIONS:
Locations (1):
- October 6 University Hospital, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided